CLINICAL TRIAL: NCT01046591
Title: Sleep and Neurobehavioral Performance After Cleft Palate Repair
Brief Title: Sleep and Behavior in Children With Cleft Palate
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Louise O'Brien, Associate Professor, University of Michigan
Other Study IDs: R000041; 1R21HL087819-01A2 (NIH)
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Cleft Palate
Keywords: Cleft Palate; Cleft Lip; Obstructive Sleep Apnea; Sleep-Disordered Breathing; Behavior; Learning
MeSH Terms: conditions — Cleft Palate; Cleft Lip; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cleft: Those with a repaired cleft palate
  Interventions: Procedure: Polysomnography
- Comparison: Those without a cleft palate repair
  Interventions: Procedure: Polysomnography

INTERVENTIONS:
Procedure: Polysomnography — Overnight sleep studies will be performed on all children.
  Other Names: PSG; Overnight polysomnography

SUMMARY:
The purpose of this study is to determine whether cleft palate repair increases the risk for obstructive sleep apnea in children and whether sleep apnea could explain learning and behavior difficulties that are often observed.

ELIGIBILITY:
Inclusion Criteria:

* Previous cleft palate repair
* Age 6-15 years

Exclusion Criteria:

* Other condition that impacts the interpretation of PSG or neurobehavioral assessments
* Being treated for sleep apnea with CPAP

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children will be recruited from cleft palate clinics
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2006-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Severity of obstructive sleep apnea | Within 24 hours of enrollment.

SECONDARY OUTCOMES:
Hyperactivity scores | Within 24 hours of enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Louise M O'Brien, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States